CLINICAL TRIAL: NCT02467153
Title: Influence of Combined Vitamin D Supplementation and Resistance Exercise Training on Musculoskeletal Health in Frail Older Men and Women (EXVITD)
Brief Title: Vitamin D and Resistance Exercise Training; Effects on Musculoskeletal Health in Frail Older Men and Women
Acronym: EXVITD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: University Hospital Birmingham (Other); University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RG_14-185
Record Dates: First submitted 2015-05-11; First posted 2015-06-09 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2021-03

CONDITIONS: Sarcopenia; Muscle Atrophy; Osteoporosis
Keywords: Sarcopenia; Older adult; Vitamin D; Physical activity; Muscle atrophy; Muscle strength; Physical function; Frailty; Osteoporosis
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy; Osteoporosis; Motor Activity; Frailty | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RET + vitamin D3 (Experimental): Resistance Exercise Training (RET) + vitamin D3 given orally as tablets at a dosage of 800 International Units (IU)/day for 6 months.
  Interventions: Other: RET; Dietary Supplement: Vitamin D3
- RET + placebo (Placebo Comparator): Resistance Exercise Training (RET) + placebo given orally as tablets; 1 tablet per day for 6 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Other: RET — RET: A supervised group exercise programme with a maximum of n=10-12 participants per group to be attended 3 times per week for 6 months.
  The RET programme includes elements of current established programmes for falls prevention/ core stability (i.e., OTAGO, PEPPI) and will tailored to a range of abilities within the target group.
  Vitamin D3 supplementation: vitamin D3 given orally as tablets at a dosage of 800 IU/day for 6 months.
  Arms: RET + vitamin D3
Dietary Supplement: Placebo — Placebo given orally as tablets; 1 tablet per day for 6 months.
  Arms: RET + placebo
Dietary Supplement: Vitamin D3 — Placebo given orally as tablets; 800 IU as 1 tablet per day for 6 months.
  Arms: RET + vitamin D3

SUMMARY:
This study aims to determine whether vitamin D3 supplementation is any more effective in improving musculoskeletal function when combined with exercise training compared with exercise training alone.

DETAILED DESCRIPTION:
We are an ageing population with life expectancy currently increasing at 2 years per decade. Crucially, healthy life expectancy is not keeping pace and older adults are now spending longer in poor health.

Sarcopenia represents a major, serious and increasing public health problem. While the causes of sarcopenia are still unclear, vitamin D deficiency, which is widespread among older adults (reaching 90% in residential care), is associated with an increased risk of falls and fractures as well as skeletal muscle weakness. While it is known that vitamin D is essential for bone health, relatively little is known about the direct effects of vitamin D3 supplementation on human muscle mass and function in humans.

Physical activity (resistance exercise training (RET) in particular) is the most potent stimulus for skeletal muscle hypertrophy in both young and older adults. The researchers and others have shown that even in very old adults (>75 years) and frail patient groups, RET improves muscle strength and functional outcomes although the hypertrophic ability of older muscle is blunted compared with younger adults. Therefore in order to help older adults maintain good musculoskeletal health, interventions to optimise responsiveness to physical activity are likely to be most effective if they are multimodal, and include resistance exercise. One example of this is to combine resistance exercise training with vitamin D supplementation.

The aim of the EXVITD study is to determine whether vitamin D3 supplementation is any more effective in improving musculoskeletal function when combined with exercise training compared with exercise training alone.

The researchers aim to recruit 127 men and women aged 65 years or over who are ambulatory (with or without walking aids) and live in supported housing settings. Recruitment will be via local housing trusts/seniors groups.

Participants will be randomised to RET (x3 per week) + 800 International Units (IU) vitamin D3 (daily) supplement or RET + placebo for six months. Participants will be stratified on the basis of vitamin D status, physical activity (measured directly pre-randomisation using accelerometry), and sex.

Tests will include, but are not limited to, lower limb extensor power (LLEP) output, body composition, Short Physical Performance Battery (SPPB), Timed-up-and-go (TUG),power required to rise from a chair, physical activity, perception of musculoskeletal comfort/pain, falls as events, quality of life and venepuncture for biochemical markers.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or over
* Ambulatory (with or without walking aids)

Exclusion Criteria:

* History of myocardial infarction within previous 2 years
* Cardiac illness: moderate/ severe aortic stenosis, acute pericarditis, acute myocarditis, aneurysm, severe angina, clinically significant valvular disease, uncontrolled dysrhythmia, claudication within the previous 10 years; thrombophlebitis or pulmonary embolus within the previous 2 years
* History of cerebrovascular disease (CVA or TIA) within the previous 2 years
* Acute febrile illness within the previous 3 months
* Severe airflow obstruction; uncontrolled metabolic disease (e.g., thyroid disease or cancer)
* Significant emotional distress, psychotic illness or depression within the previous 2 years
* Lower limb fracture sustained within the previous 2 years/ upper limb fracture within the previous 6 months
* Non-arthroscopic lower limb joint surgery within the previous 2 years
* Any reason for loss of mobility for greater than 1 week in the previous 2 months or greater than 2 weeks in the previous 6 months
* Resting systolic pressure >200 millimeters of mercury (mmHg) or resting diastolic pressure >100 mmHg
* Poorly controlled atrial fibrillation; poor (chronic) pain control
* Moderate/severe cognitive impairment (mini mental state examination (MMSE) score <23)
* Vitamin D deficient (serum 25(OH)D3 <30nmol/l); current antiresorptive or anabolic treatment for osteoporosis
* Treatment with bisphosphonates for osteoporosis in the past two years
* Current supplement use of vitamin D (>400 IU/day) or calcium (>500 mg/day including use of over the counter preparations)
* Current use of glucocorticoids; known primary hyperparathyroidism; hypercalcaemia (albumin-adjusted serum calcium >2.60 mmol/l)
* Renal impairment (Stage 4 or 5)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Lower limb extensor power (LLEP) | 6 months
  Nottingham Leg Extensor Power Rig

SECONDARY OUTCOMES:
Body composition and bone mineral density (BMD) | 6 months
  Body composition, hip and spine BMD measured using dual-energy X-ray absorptiometry (DXA)
Short Physical Performance Battery (SPPB) | 6 months
  Gait speed, chair stand, balance tests
Timed-up-and-go (TUG) | 6 months
  To assess mobility
Physical activity | 6 months
  Directly monitored physical activity using accelerometry (ActivPAL)
Falls as events | 6 months
  Incidence of falls
Quality of life (QoL) | 6 months
  QoL assessed via questionnaire
Serum blood monitoring | 6 months
  Venepuncture for markers of inflammation plus monitoring of serum vitamin D3 and calcium status at baseline, 1, 3 and 6 months.
Muscle power | 6 months
  Chair rise test using Leonardo Mechanograph Ground Reaction Force Plate
3-day Dietary analysis | 6 months
  3-day food diary record

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Greig, PhD, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, United Kingdom

REFERENCES:
- [Derived] Welford AE, Lanham-New S, Lord J, Doyle A, Robinson J, Nightingale P, Gittoes N, Greig CA. Influence of combined vitamin D3 supplementation and resistance exercise training on musculoskeletal health in older men and women (EXVITD): protocol for a randomised controlled trial. BMJ Open. 2020 Mar 18;10(3):e033824. doi: 10.1136/bmjopen-2019-033824. PMID 32193264